CLINICAL TRIAL: NCT00546481
Title: An Open-label, Randomized, Multi-center, Parallel Group Study to Demonstrate Correction of Anemia Using Intravenous Injections of RO0503821 in Patients With Chronic Kidney Disease Who Are on Dialysis
Brief Title: A Study of Intravenous Mircera for the Correction of Anemia in Dialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20884
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Erythropoietin

ARMS (2):
- Correction Phase: CERA (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [RO0503821, Mircera]
- Correction Phase: Epoetin Beta (Active Comparator)
  Interventions: Drug: Epoetin

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [RO0503821, Mircera] — 0.6 micrograms/kg every 2 weeks
  Arms: Correction Phase: CERA
Drug: Epoetin — As prescribed, iv, 3 times weekly
  Arms: Correction Phase: Epoetin Beta

SUMMARY:
This 2 arm study will evaluate the efficacy of intravenous Mircera treatment for the correction of anemia in patients with chronic kidney disease who are on dialysis. Patients will be randomized to receive either Mircera 0.6 micrograms/kg i.v. every 2 weeks, or epoetin 3 times per week i.v. according to approved treatment recommendations. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* maintenance hemodialysis or peritoneal dialysis for >=2 weeks before screening, and during screening period.

Exclusion Criteria:

* previous therapy with epoetin within 8 weeks prior to screening;
* overt gastrointestinal bleeding within 8 weeks before screening or during screening period;
* RBC transfusions within 8 weeks before screening or during screening period;
* active malignant disease except non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- South Korea (3):
  - Gyeonggi-do
  - Seoul
  - Sungnam

REFERENCES:
- [Derived] Oh J, Joo KW, Chin HJ, Chae DW, Kim SG, Kim SJ, Chung W, Kim S, Huh W, Oh HY, Choi BS, Yang CW, Kim S. Correction of anemia with continuous erythropoietin receptor activator in Korean patients on long-term hemodialysis. J Korean Med Sci. 2014 Jan;29(1):76-83. doi: 10.3346/jkms.2014.29.1.76. Epub 2013 Dec 26. PMID 24431909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were enrolled in this study conducted from 05 November 2007 to 23 December 2009 at 7 centers in Korea.
Groups:
- Correction Phase: CERA: Eligible participants were administered CERA IV once every 2 weeks at the starting dose of 0.6 μg/kg for 24 weeks.
- Correction Phase: Epoetin Beta: Eligible participants were administered Epoetin beta IV three times per week at the starting dose of 40 IU/kg for 24 weeks.
- Maintenance Phase: CERA: Eligible participants who achieved a hemoglobin target range of level >=11.0 g/dL at least once during the correction phase (Week 1 to Week 24) without RBC transfusion and completed correction phase treatment, moved to Maintenance phase wherein they were administered CERA (dose adjusted according to the predefined criteria in protocol) IV once every 4 weeks for the subsequent 24 weeks.
Period: Correction Phase (CERA or Epoetin Beta)
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Maintenance Phase: CERA
Started | 39 | 41 | 0
Completed | 33 | 36 | 0
Not Completed | 6 | 5 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Kidney transplantation | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — RBC transfusion | 0 | 1 | 0
Period: Maintenance Phase (CERA)
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Maintenance Phase: CERA
Started | 0 | 0 | 54
Completed | 0 | 0 | 50
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Kidney transplantation | 0 | 0 | 1
Not completed — Other Reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (15.3) | 54.3 (12.8) | 54.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hemoglobin Response up to Week 24
Description: Hemoglobin (Hb) response was defined as increase of Hb by at least 1 g/dL compared with baseline and Hb>/=11 g/dL without red blood cell transfusion during 24-week correction phase. The average baseline value was estimated by the mean of all values recorded between the day of first study dose and the previous 20 days. The percentage of participants who achieved Hb response is presented
Time Frame: Up to Week 24
Population: The Intent-to-Treat population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 39 | 41
Percentage of participants | 79.5 [63.5 to 90.7] | 87.8 [73.8 to 95.9]

2. Secondary Outcome: Mean Change From Baseline in Hemoglobin Concentration at Week 24
Description: Mean hemoglobin levels and their changes in correction phase from baseline were presented. Baseline is defined as Day 1 visit. The mean Hb concentration from Baseline at week 24 was calculated by subtracting the baseline Hb concentration value from the week 24 value
Time Frame: From Baseline (Day 1) to Week 24
Population: The Intent-to-Treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 39 | 41
Grams per deciliter (g/dL) | 2.00 (1.51) | 2.03 (1.37)

3. Secondary Outcome: Median Time in Which Hemoglobin Value Was Maintained Within Target Range of >/= 11g/dL up to Week 24
Description: Median time during the correction period in which Hb value was maintained within target range of >/= 11.0 g/dL and an increase in hemoglobin from baseline >/= 1.0 g/dL was reported.
Time Frame: Up to Week 24
Population: The Intent-to-Treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 39 | 41
Days | 84 [70 to 98] | 72 [58 to 72]

4. Secondary Outcome: Number of Participants Who Received Red Blood Cells Transfusions up to Week 49
Description: The number of participants who received at least 1 red blood cell transfusion during the study is presented. RBC transfusions was given in case of medical need, i.e., in severely anemic participants with recognized symptoms or signs of anemia (e.g., in participants with acute blood loss, with severe angina, or whose Hb decreases to critical levels)
Time Frame: Up to Week 49
Population: The Intent-to-Treat Population included all randomized participants.
Measure: Number; unit: Number of participants
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Maintenance Phase: CERA
Number analyzed (Participants) | 39 | 41 | 54
Number of participants | 8 | 2 | 1

5. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Number of participants with at least one AE and SAE were reported.
Time Frame: Up to Week 49
Population: All participants who received at least one dose of the study medication and had a safety follow-up, whether withdrawn prematurely or not, included in the Safety Population. One participant from CERA group and two participants from Epoetin Beta group did not receive any study medication and were excluded from the safety analysis.
Measure: Number; unit: Number of participants
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Maintenance Phase: CERA
Number analyzed (Participants) | 38 | 39 | 54
Number of participants
  Number of participants with any AE | 34 | 39 | 51
  Number of participants with any SAE | 10 | 6 | 8

6. Secondary Outcome: Mean Change From Baseline in Vital Signs: Systolic Blood Pressure and Diastolic Blood Pressure up to Week 24
Description: Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Baseline and end of correction phase (Week 24) is presented. SBP and DBP were determined both before and after the dialysis session for participants. Baseline is defined as Day 1 visit. One participant from CERA group and two participants from Epoetin Beta group did not receive any study medication and were excluded from the safety analysis.
Time Frame: From Baseline (Day 1) to Week 24
Population: All participants who received at least one dose of the study medication and had a safety follow-up, whether withdrawn prematurely or not, included in the Safety Population. Only participants available at the time of assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 38 | 39
millimeters of mercury
  Pre-dialysis: SBP | 2.74 (22.5) | 2.72 (19.2)
  Pre-dialysis: DBP | -1.74 (13.3) | 3.87 (11.5)
  Post-dialysis: SBP | 5.26 (22.3) | 2.59 (23)
  Post-dialysis: DBP | 0.84 (13.7) | 3.28 (11.7)

7. Secondary Outcome: Mean Change From Baseline in Vital Sign: Heart Rate Measurements up to Week 24
Description: Heart rate was measured before blood sampling for all participants and before the dialysis session. Baseline is defined as Day 1. One participant from CERA group and two participants from Epoetin Beta group did not receive any study medication and were excluded from the safety analysis.
Time Frame: From Baseline (Day 1) to Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute for heart rate
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 38 | 39
Beats per minute for heart rate | -5.39 (13.5) | -1.79 (10.1)

8. Secondary Outcome: Number of Participants With Abnormal Changes in Electrocardiogram up to Week 24
Description: Twelve-lead ECG was recorded before or after the dialysis session. Number of participants with abnormal changes in electrocardiogram observed at any time point was reported. One participant from CERA group and two participants from Epoetin Beta group did not receive any study medication and were excluded from the safety analysis.
Time Frame: Up to Week 24
Population: as for outcome 6
Measure: Number; unit: Number of participants
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta
Number analyzed (Participants) | 36 | 32
Number of participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to Week 49
Description: All participants who received at least one dose of the study medication and had a safety follow-up, whether withdrawn prematurely or not, included in the Safety Population. One participant from CERA group and two participants from Epoetin Beta group did not receive any study medication and were excluded from the safety analysis.
Groups:
- Maintenance Phase: CERA: Eligible participants who achieved a hemoglobin target range of level >=11.0 g/dL at least once during the correction phase (Week 1 to Week 24) without RBC transfusion and completed correction phase treatment, moved to Maintenance phase wherein they were administered CERA (dose adjusted according to the predefined protocol) IV once every 4 weeks for the subsequent 24 weeks.
Arm/Group | Correction Phase: CERA | Correction Phase: Epoetin Beta | Maintenance Phase: CERA
Serious Adverse Events (participants affected / at risk) | 10/38 | 6/39 | 8/54
Other Adverse Events (participants affected / at risk) | 34/38 | 39/39 | 51/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Correction Phase: CERA (N=38) | Correction Phase: Epoetin Beta (N=39) | Maintenance Phase: CERA (N=54)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Meniscus lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1 | 0
Stupor (Nervous system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Reocclusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Correction Phase: CERA (N=38) | Correction Phase: Epoetin Beta (N=39) | Maintenance Phase: CERA (N=54)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 4
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 5
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3
Chest discomfort (General disorders) | 3 | 2 | 3
Chest pain (General disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 14 | 9
Upper respiratory tract infection (Infections and infestations) | 9 | 10 | 16
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 4 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Haemodialysis - induced symptom (Injury, poisoning and procedural complications) | 3 | 3 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 6 | 4 | 6
Vascular graft complication (Injury, poisoning and procedural complications) | 3 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 3 | 6
Blood phosphorus increased (Investigations) | 1 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 6 | 2 | 5
Paraesthesia (Nervous system disorders) | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 4
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Renal cyst (Renal and urinary disorders) | 2 | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Tooth extraction (Surgical and medical procedures) | 2 | 0 | 0
Hypertension (Vascular disorders) | 6 | 2 | 5
Hypotension (Vascular disorders) | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.